CLINICAL TRIAL: NCT03711110
Title: Cardiotoxicity in the Elderly. Comparative Clinical Trial Between Primary Versus Secondary Cardiovascular Prevention Strategies
Brief Title: Cardiovascular Prevention Strategies in Elderly Patients With Cancer (CARTIER Clinical Trial)
Acronym: CARTIER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León (Other)
Collaborators: Instituto de Investigación Biomédica de Salamanca (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CARTIER
Record Dates: First submitted 2018-10-09; First posted 2018-10-18 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Cancer (Colon Cancer, Breast Cancer, Lymphoma, Chronic Lymphoma Leukemia, Multiple Myeloma); Elderly; Antineoplastic Agents; Cardiotoxicity
Keywords: Cardiotoxicity; Elderly; Antineoplastic agents; Cardiovascular monitoring; Cardioprotection; Cardio-oncology; Chemically-Induced Disorders; Radiation Injuries; Drug-Related Side Effects and Adverse Reactions.; Primary prevention; Secondary prevention.; Mortality
MeSH Terms: conditions — Neoplasms; Colonic Neoplasms; Breast Neoplasms; Lymphoma; Multiple Myeloma; Cardiotoxicity; Chemically-Induced Disorders; Radiation Injuries; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Intervention Model Description: Randomized, multicenter, open-label clinical trial comparing, in elderly patient with cancer under anti-tumoral treatment, two different cardiotoxicity prevention strategies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary prevention strategy (Experimental): Intensive cardiovascular monitoring focused on prevention and early diagnosis and treatment of cardiotoxicity based in cardio-onco-hematology teams involved in cancer patient care.
  Interventions: Other: Intensive cardiovascular monitoring
- Secondary prevention strategy (control) (Other): Current clinical practice: cardiac care is based on the onco-hematologist criteria.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Intensive cardiovascular monitoring — Schedule of visits: Evaluation before starting chemotherapy, at three and six months and annually for five years (eight visits: baseline, 3rd and 6th month, 1st, 2nd, 3rd, 4th and 5th years).
  Assessment protocol: Anamnesis and physical examination; EKG; Echocardiogram; Biomarkers (troponin and natriuretic peptide); Structured counselling on healthy cardiac practices; Treatment optimization of cardiovascular risk factors and heart diseases; Quality of life (ECOG Performance status and Minnesota questionnaires); Interaction and management of patient care by the cardio-onco-hematology team. Moreover, cardiac MRI in centers participating in the CARTIER-MR sub-study.
  Arms: Primary prevention strategy
Other: No intervention — Schedule of visits: Evaluation before starting chemotherapy, at three and six months and annually for five years (eight visits: baseline, 3rd and 6th month, 1st, 2nd, 3rd, 4th and 5th years).
  Assessment protocol: Anamnesis and physical examination; ECOG Performance status; cardiac patient care based on the onco-hematologist criteria
  Arms: Secondary prevention strategy (control)

SUMMARY:
The CARTIER study is a randomized, multicenter, open-label clinical trial comparing, in elderly patients with cancer under anti-tumoral treatment, two different cardiotoxicity prevention strategies: primary (intensive cardiovascular monitoring focused on prevention and early diagnosis and treatment of cardiotoxicity based in cardio-onco-hematology teams involved in cancer patient care) vs. secondary (current clinical practice where intensive cardiovascular monitoring is not routinely performed and cardiotoxicity patient care is based on the onco-hematologist criteria).

The primary endpoint is to determine whether this primary prevention englobing cardiovascular monitoring plus intensive multidisciplinary management is superior to the current clinical practice in reducing all cause mortality.

Other secondary objectives of the study are to analyze the impact of this intensive cardiovascular monitoring strategy on the incidence of cardiovascular mortality, oncological mortality, hospitalization and/or urgent care due to cardiovascular complications, hospitalization and/or urgent oncological care due to cancer complications, tumor progression and cost-effectiveness analysis.

A total of 514 patients ≥ 65 years old diagnosed with any of the following onco-hematological cancers, colon, breast, lymphoma, chronic lymphoma leukemia, chronic myeloid leukemia or myeloma, undergoing standardized anti-tumoral treatment, will be recruited.

The incidence of primary and secondary outcomes will be measured at 2 and 5 years

ELIGIBILITY:
Inclusion Criteria:

* > 65 years old
* Expected survival >1 year
* Colon cancer, breast cancer, lymphoma, chronic lymphoma leukemia, chronic myeloid leukemia, myeloma
* Signature on the informed consent

Exclusion Criteria:

* Patients included in clinical trials will be excluded if they interfere with the CARTIER follow-up protocol. If they do not interfere they can be included
* Patients who had received previous potentially cardiotoxic anticancer treatment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 514 (Estimated)
Dates: Start 2019-08-02 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | Two (mid-term analysis) and five years of follow-up
  Cumulative incidence of all-cause mortality

SECONDARY OUTCOMES:
Oncological mortality | Two and five years of follow-up
  Cumulative incidence of oncological mortality
Cardiovascular mortality | Two and five years of follow-up
  Cumulative incidence of cardiovascular mortality
Hospitalization | Two and five years of follow-up
  Cumulative incidence of hospitalization
Hospitalization/emergency cardiovascular cause | Two and five years of follow-up
  Cumulative incidence of hospitalization and/or emergency care for cardiovascular cause
Hospitalization/emergency cancer cause | Two and five years of follow-up
  Cumulative incidence of hospitalization and/or emergency care for cancer cause
Tumor recurrence or progression | Two and five years of follow-up
  Incidence of tumoral recurrence or progression

CONTACTS AND LOCATIONS:
Overall Officials: Pedro L Sánchez, Ph. D., Study Director — IBSAL-Instituto de Investigación Biomédica de Salamanca; Ana Martín-García, Ph. D., Study Director — IBSAL-Instituto de Investigación Biomédica de Salamanca
Locations (14):
- Spain (14):
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Hospital de Galdakao-Usansolo, Galdakao, Vizcaya
  - Hospital Universitario Vall d´Hebron, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario de La Princesa, Madrid
  - Hospital G. Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Río Hortega, Valladolid